CLINICAL TRIAL: NCT04737395
Title: Intensive Upper Extremity Training Program During the Early Subacute Phase After Stroke: A Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Aleh Negev Nahalat Eran, Israel (Unknown); Ben-Gurion University of the Negev, Israel (Unknown)
Responsible Party: Principal Investigator, Dr. Oren Barzel, Director of the Orthopedic Rehabilitation Department, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-19-6218-OB-CTIL
Record Dates: First submitted 2021-01-19; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Device-assisted therapy ("Meditouch","MSQUARE") (Experimental): 40 hours of therapy with the the Hand Tutor (MediTouch) device and a wearable vest (MSQUARE) for arm rehabilitation
  Interventions: Device: upper extremity training program ("Meditouch","MSQUARE")

INTERVENTIONS:
Device: upper extremity training program ("Meditouch","MSQUARE") — 40 hours of therapy with the Hand Tutor (MediTouch) device and a wearable vest (EkssoUE, Ekso Bionics) for arm rehabilitation

SUMMARY:
The study assesses the feasibility of a 4-week upper extremity training program emphasizing quality of movement practiced at high intensity and dosage applied during the early subacute phase after stroke.

DETAILED DESCRIPTION:
Participants will receive 120 minutes of upper extremity training X 5 days per week for 4 weeks in addition to their daily rehabilitative routine (total therapy time 40 hours in addition to daily routine treatments of approximately 60 hours). Each session will be staffed with a 1:1 PT/OT to patient ratio.

The aim of the program is to increase the time spent on tasks using customized game-based platforms that include highly immersive, challenging and rewarding virtual environments for upper limb training. The focus of these game-based platforms is to reduce upper extremity impairments through emphasizing the quality of movement execution.

In one platform, the participant controls virtual dolphin movements by moving his/her paretic upper limb. The game utilizes advanced artificial intelligence (AI) analysis of the video recordings in real-time. In case the participant needs arm weight support, the practice will perform the task with a mechanical wearable exoskeleton vest, EkssoUE (Ekso Bionics) that can provide support at different weight levels. Arm weight support will be titrated as the patient progresses through each session and will be reduced/removed if no significant compensatory strategies were used.

The second platform, the HandTutor system (MediTouch) consists of an ergonomic wearable glove and a dedicated software with games that allow practicing active wrist movements, grip control and finger individuation in a challenging and motivating environment. Participant progresses through simple to difficult games while adjusting the range of motion that is being practiced according to participant's abilities.

Training in both platforms will be conducted in sitting. Participant will continue with their regular rehabilitative routine that includes daily physical and occupational therapy sessions and speech therapy if needed as well as group work and gym.

To assess the feasibility of the proposed intervention the following data/measures will be documented:

Adherence rates; Time on task (in minutes); Progression in game levels and the amount of weight support; Attendance to routine rehabilitative sessions; Visual Analogue Scale will be used to monitor the levels of pain; Rating perceived exertion (RPE), the revised category-ratio scale (0 to 10 scale) will be used to monitor and guide exercise intensity; The Pittsburgh rehabilitation participation scale (PRPS); The Intrinsic Motivation Inventory (IMI) - will be assessed at the end of intervention period; Acceptability and satisfaction of the intervention to participants will be assessed at the end of training period using a self-designed questionnaire/rating scale; Adverse events; Problems/difficulties related to intervention equipment (software, hardware, vest etc.).

To evaluate the potential effectiveness of the intervention the following data/measures will be conducted at baseline (prior training), immediately post intervention and at 12 (±14) and 24 (±14) weeks post stroke:

Fugl-Meyer upper extremity assessment (FM-UE); Action research arm test (ARAT); Stroke Impact Scale (SIS) hand domain, version 2.0; Upper extremity impairment and function will be assessed using a reaching and a grasping tasks that will be recorded using multiple high resolution video-cameras and analyzed using AI algorithm (OpenPose).

ELIGIBILITY:
Inclusion criteria:

* age ≥18 years;
* Ischemic or hemorrhagic stroke (hemispheric or brainstem) confirmed by CT or MRI;
* First-ever stroke or previous stroke with no upper extremity weakness;
* 1 week ≤ Time after stroke onset ≤ 6 weeks;
* Active shoulder flexion of at least 20◦ and partial wrist and/or finger active movement;
* Ability to provide inform consent.

Exclusion criteria:

* A painful shoulder limiting an active forward reach;
* Severe spasticity or non-neural loss of range of motion;
* Cognitive or communication impairments as determined by the clinical team;
* Unstable medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-22 (Actual); Primary Completion 2022-11-22 (Estimated); Study Completion 2022-11-22 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer upper extremity assessment (FM-UE) | From baseline to day 3 post-training
  Change in arm impairment, measured by FM-UE. Maximum score (Performs fully) =226 points Minimum score= 0 points

SECONDARY OUTCOMES:
Action research arm test (ARAT) | From baseline to day 3 post-training
  Change in arm function, measured by. Maximum score (Performs fully) = 57 points Minimum score= 0 points
Stroke Impact Scale (SIS) | From baseline to day 3 post-training
  Change in disability and health related quality of life Maximum score (Performs fully) = 25 points Minimum score= 0 points

CONTACTS AND LOCATIONS:
Locations (1):
- Aleh Negev Nahalat Eran, Ofakim, Israel

IPD SHARING:
Plan to Share IPD: No